CLINICAL TRIAL: NCT00185523
Title: Allogeneic Peripheral Blood Stem Cell Transplantation for Patients With Acute Myelogenous Leukemia and Acute Lymphoblastic Leukemia in First or Second Remission or Chronic Myelogenous Leukemia in First and Second Chronic Phase or Accelerated Phase
Brief Title: Allogeneic Transplantation for Patients With Acute Leukemia or Chronic Myelogenous Leukemia (CML)
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: BMT142; 78149; NCT00185523; 12570 (Other: Stanford IRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia, Lymphocytic, Acute; Leukemia; Leukemia Acute Promyelocytic Leukemia (APL); Leukemia Acute Lymphoid Leukemia (ALL); Leukemia Chronic Myelogenous Leukemia (CML); Leukemia Acute Myeloid Leukemia (AML); Leukemia Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Leukemia, Promyelocytic, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- CML in first Chronic Phase or Accelerated Phase: Busulfan/cyclophosphamide Day -7: Busulfan 1.0 mg/kg IV q6 hrs** Day -6: Busulfan 1.0 mg/kg IV q6 hrs Day -5: Busulfan 1.0 mg/kg IV q6 hrs Day -4: Busulfan 1.0 mg/kg IV q6 hrs Day -3: Cyclophosphamide 60 mg/kg Day -2: Cyclophosphamide 60 mg/kg Day -1: rest Day 0: Allogeneic PBSC infusion
  Interventions: Procedure: Allogeneic hematopoietic cell transplantation
- AML and ALL in first or second remission: FTBI/VP-16 Day -7: FTBI 120 cGy x 3 fractions Day -6: FTBI 120 cGy x 2 fractions Day -5: FTBI 120 cGy x 3 fractions Day -4: FTBI 120 cGy x 3 fractions* Day -3: VP-16 at 60 mg/kg Day -2: rest Day -1: rest Day 0: Allogeneic PBSC infusion
  Interventions: Procedure: Allogeneic hematopoietic cell transplantation

INTERVENTIONS:
Procedure: Allogeneic hematopoietic cell transplantation

SUMMARY:
The purpose of the study is to evaluate the overall and disease free survival of recipients who have received G-CSF mobilized stem cells from HLA matched sibling donors.

DETAILED DESCRIPTION:
Allogeneic Peripheral Blood Stem Cell Transplantation for Patients with Acute Myelogenous Leukemia and Acute Lymphoblastic Leukemia in First Remission or Chronic Myelogenous Leukemia in First Chronic Phase

ELIGIBILITY:
Inclusion Criteria:1. Any patient with one of the following hematologic malignancies in whom an allogeneic stem cell transplant is warranted: Specific disease categories include:

1. acute myelogenous leukemia, 1st or 2nd remission
2. acute lymphoblastic leukemia, 1st or 2nd remission
3. chronic myelogenous leukemia, 1st or 2nd CP, accelerated phase 2. Patient age > 1 month and < 55 yo 3. Patients must have a genotypically HLA identical sibling 4. Patient must have adequate function as follows:

a. total bilirubin <2.5 and SGOT/SGPT <2x normal b. adequate renal function as defined by creatinine < 1.5 or a 24 hr creatinine clearance >50 cc/min as determined by the Cockroft-Gault formula (to be done if serum creatinine > 1.5) c. DLCO > 60% predicted d. radionuclide cardiac scan with ejection fraction >45% 5. Patient must be competent to give consent.

Inclusion criteria (Donor):

1. HLA identical family member
2. Donor or guardian must be competent to give consent
3. Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter

Exclusion Criteria:3.2 Exclusion Criteria (Patient):

1. Evidence of active infection or active hepatitis
2. Positive serologies for HIV-1,HIV-2 or hepatitis B surface ag+
3. Previous allogeneic stem cell/bone marrow transplant
4. Pregnant or lactating patients

4 Exclusion criteria (Donor):

1. Donors who for psychologic, physiologic or medical reasons are unable to tolerate PBSC harvest
2. Donors who are HIV+ or hepatitis B antigen +
3. History of allergic reaction to G-CSF
4. Female donors must be post-menopausal or have a negative pregnancy test

Ages: 4 Weeks to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2002-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall and disease free survival of recipients who have received G-CSF mobilized stemcells from their donors. | no known

CONTACTS AND LOCATIONS:
Overall Officials: Ginna Laport, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States